

| THE PARENT/LEGAL GUARDIAN AND CHILD |
|---|
| (Name and surname of the parent/legal guardian of the child) |
| (Contact details: e-mail address, postal address, and phone number) |
| In accordance with Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natural persons regarding the processing of personal data and on the free movement of such data, and repealing Directive 95/46/EC (General Data Protection Regulation, hereinafter referred to as GDPR), and the Act of 10 May 2018 on the Protection of Personal Data – I consent to the processing of my personal data and the personal data of my child: |

(Name and surname, residential address, date of birth, and PESEL number of the child – study participant)

by the Medical University of Gdańsk for the purpose of conducting the study entitled "Evaluation of the Effectiveness of Functional Constipation Treatment", in which the child will participate, as well as the potential sharing of the above data with entities authorized by law.

- 1. The scope of processed personal data includes: full name, date of birth, PESEL number, residential address, correspondence address, telephone number, and e-mail address.
- 2. Providing consent for the processing of the personal data of the parent/legal guardian and the child is voluntary.
- 3. Personal data will be obtained from the parents/legal guardians of the child based on this declaration (Art. 6(1)(a) and Art. 9(2)(j) GDPR).
- 4. The data controller is the Medical University of Gdańsk, located at ul. M. Skłodowskiej-Curie 3a, 80-210 Gdańsk, represented by the Rector.



- 5. The data controller has appointed a Data Protection Officer who can be contacted regarding personal data processing via email at <a href="mailto:iod@gumed.edu.pl">iod@gumed.edu.pl</a> or by phone at +48 58 349 10 27.
- 6. The data controller does not disclose personal data to any recipients unless required by generally applicable law or an agreement entered into by the controller.
- 7. The data will be stored for the duration of the study and until the study results are developed and utilized.
- 8. The parent/legal guardian has the right to access their own and the child's personal data, to rectify, erase, or restrict its processing.
- 9. The parent/legal guardian has the right to object to further processing and to withdraw consent to the continued processing of their own and the child's personal data. The withdrawal of consent does not affect the legality of processing carried out prior to its withdrawal.
- 10. The parent/legal guardian has the right to data portability regarding their own and the child's personal data.
- 11. The parent/legal guardian has the right to lodge a complaint regarding the processing of their own and the child's personal data by the controller with the President of the Personal Data Protection Office.

| (Date and legible signature of the parent/legal guardian of the child) |
|------------------------------------------------------------------------|
| (Date and legible signature of the study participant)* |
| *To be filled in if the study participant is over 13 years of age. |



## OŚWIADCZENIE O WYRAŻENIU ZGODY NA PRZETWARZANIE DANYCH OSOBOWYCH WŁASNYCH I DZIECKA

| (Imię i nazwisko rodzica/opiekuna prawnego dziecka) |
|---|
| (Dane kontaktowe: adres e-mail, adres korespondencyjny i numer telefonu) |
| Zgodnie z Rozporządzeniem Parlamentu Europejskiego i Rady (UE) 2016/679 z dnic 27.04.2016r. w sprawie ochrony osób fizycznych w związku z przetwarzaniem danycł osobowych i w sprawie swobodnego przepływu takich danych oraz uchylenic dyrektywy 95/46/WE (ogólne rozporządzenie o ochronie danych) Dz. Urz. UE L z 2016/nr 119/1- (zwanym dalej RODO) oraz ustawy z dnia 10.05.2018 r. O ochronie danycł osobowych - wyrażam zgodę na przetwarzanie moich danych osobowych i danycł osobowych mojego dziecka: |
| (Imie i nazwisko, adres zamieszkania, data urodzenia oraz PESEL dziecka-uczestnika hadania) |

przez Gdański Uniwersytet Medyczny w celu realizacji badania "Ocena skuteczności leczenia zaparć czynnościowych", w którym dziecko będzie uczestniczyło oraz ewentualnego udostępnienia przedmiotowych danych uprawnionym z mocy prawa podmiotom.

- 1. Zakres przetwarzanych danych osobowych obejmuje: imię i nazwisko, data urodzenia, PESEL, adres zamieszkania, adres korespondencyjny, telefon, adres email.
- 2. Udzielenie zgody na przetwarzanie danych osobowych rodzica/opiekuna prawnego i dziecka jest dobrowolne.
- 3. Dane osobowe będą pozyskiwane od rodziców/opiekunów prawnych dziecka, na podstawie niniejszego oświadczenia (art. 6 ust. 1 lit. a art. 9 ust. 2 lit. j RODO).



- 4. Administratorem danych osobowych jest Gdański Uniwersytet Medyczny z siedzibą przy ul. M. Skłodowskiej-Curie 3a, 80-210 Gdańsk, reprezentowany przez Rektora.
- 5. Administrator wyznaczył Inspektora Ochrony Danych, z którym można kontaktować się w sprawach dotyczących przetwarzania danych osobowych pod adresem e-mail: <a href="mailto:iod@gumed.edu.pl">iod@gumed.edu.pl</a> lub nr tel.: 58 349 10 27.
- 6. Administrator nie udostępnia danych osobowych żadnym odbiorcom z wyjątkiem, gdy obowiązek taki wynika z przepisów prawa powszechnie obowiązującego lub umowy zawartej przez Administratora.
- 7. Dane będą przechowywane przez czas trwania badania oraz do czasu opracowania i wykorzystania jego wyników.
- 8. Rodzic/opiekun prawny ma prawo dostępu do swoich danych osobowych oraz danych osobowych dziecka, ich sprostowania, usunięcia lub ograniczenia przetwarzania.
- 9. Rodzic/opiekun prawny ma prawo do wniesienia sprzeciwu wobec dalszego przetwarzania, wycofania zgody na dalsze przetwarzanie swoich danych osobowych oraz danych osobowych dziecka. Skorzystanie z prawa wycofania zgody nie ma wpływu na przetwarzanie, które miało miejsce do momentu wycofania zgody.
- 10. Rodzic/opiekun prawny ma prawo do przenoszenia swoich danych osobowych oraz dziecka.
- 11. Rodzic/opiekun prawny ma prawo wniesienia skargi na czynności przetwarzania swoich danych osobowych oraz dziecka przez Administratora do Prezesa Urzędu Ochrony Danych Osobowych

| ıta i czytelny podpis rodzica/opiekuna prawnego dziecka) |
|----------------------------------------------------------|
| ta i czytelny podpis uczestnika badania)* |



Wypełnić jeśli uczestnik badania ma powyżej 13 lat